CLINICAL TRIAL: NCT03465774
Title: A Prospective Observational Cohort Study of Indwelling Pleural Catheters Versus Indwelling Pleural Catheters Plus Doxycycline Pleurodesis for Treatment of Malignant Pleural Effusions
Brief Title: Indwelling Pleural Catheters With or Without Doxycycline in Treating Patients With Malignant Pleural Effusions
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0973; NCI-2018-00630 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0973 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pleural Neoplasm
MeSH Terms: conditions — Pleural Neoplasms | interventions — Doxycycline; Catheters, Indwelling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 2 (IPC alone): Patients undergo IPC placement.
  Interventions: Device: Indwelling Catheter; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration
- Group I (IPC, doxycycline): Patients undergo IPC placement and receive doxycycline via IPC 5 days later.
  Interventions: Drug: Doxycycline; Device: Indwelling Catheter; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Drug: Doxycycline — Receive via IPC
  Other Names: Doxycycline Monohydrate
  Groups: Group I (IPC, doxycycline)
Device: Indwelling Catheter — Receive IPC
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This study is designed to obtain preliminary data comparing indwelling pleural catheters (IPCs) versus IPCs plus doxycycline for pleurodesis as treatments for malignant pleural effusion (MPE). Indwelling pleural catheters (IPCs) are commonly used to treat pleural effusions (build-up of fluid in the lungs). Doxycycline is an antibiotic that is also used to treat pleural effusions. The goal of this clinical research study is to learn if adding doxycycline to the use of an IPC can lead to shorter treatment times with IPCs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data comparing indwelling pleural catheters (IPCs) versus IPCs plus doxycycline for pleurodesis as treatments for malignant pleural effusion (MPE).

OUTLINE: Patients choose 1 of 2 groups.

GROUP I: Patients undergo IPC placement and receive doxycycline via IPC 5 days later.

GROUP II: Patients undergo IPC placement.

After completion of study treatment, patients are followed up at 10-14 days and then monthly for up to a year.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with MPE undergoing IPC placement
* Sufficient mental capacity to provide informed consent and answer Short-Form Six-Dimension health index (SF-6D) and Borg score questions
* Inpatients that are expected to be discharged within 5 days of receiving an indwelling pleural catheter

Exclusion Criteria:

* Patients undergoing pleurodesis for benign disease (e.g., spontaneous pneumothorax)
* Inability or unwillingness to give informed consent
* Inability to perform phone call and clinical follow-up at MD Anderson Cancer Center (MDACC)
* Pregnancy
* Previous intrapleural therapy for MPE on the same side
* Eastern Cooperative Oncology Group (ECOG) of 4 and life expectancy =< 2 weeks
* Doxycycline allergy
* Extensive loculations or hydropneumothorax or other contraindication to pleurodesis
* Chylous effusions associated with malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with MPE undergoing IPC placement
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to pleural catheter removal | Up to 1 year
  This outcome will be analyzed by cause-specific hazard Cox model with treatment group as a covariate. Whenever a catheter is removed, the cause for removal will be documented. For the analysis, causes will include removal due to decreased drainage (i.e., as per plan) as well as removal due to complications (e.g. infection, empyema, refractory pain) or other reasons (e.g. catheter plugged but no complication to the patient, patient preference without a complication). We will also analyze time to catheter removal for any cause and conduct pre-specified secondary analyses to evaluate the effect of fluid drainage amount (i.e., how much was being put out from the indwelling pleural catheter (IPC) the day of IPC placement and on the day of doxycycline instillation) and size of residual effusion as assessed by chest x-ray (CXR) (on day of IPC placement and day of doxycycline instillation) on time to catheter removal.

SECONDARY OUTCOMES:
Recurrence of effusion requiring drainage after IPC | Up to 1 year
Indwelling pleural catheters (IPC) complications | Up to 1 year
Quality-adjusted survival measured using Short-Form Six-Dimension health index (SF-6D) | Baseline up to 1 year
  Will use the Kaplan-Meier product-limit method to estimate median quality-adjusted life years (QALYs) following IPC placement.
Change in dyspnea using Borg score | Baseline up to 1 year
  Will use paired t-test to compare baseline and 1 month Borg scores and utilities. A generalized linear model will be used to evaluate whether other variables have any impact on the pairwise differences between baseline and 1 month.
Assessment of symptom burden | Baseline up to 1 year
Procedure-associated pain | Up to 1 year
Need for hospitalization due to pleurodesis pain | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Ost, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org